CLINICAL TRIAL: NCT04669262
Title: A Phase 1, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of BGB-DXP604 Alone and in Combination With BGB-DXP593 in Healthy Subjects
Brief Title: BGB-DXP604 Alone and in Combination With BGB-DXP593 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: BGB-DXP604-101
Record Dates: First submitted 2020-12-04; First posted 2020-12-16 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: BGB-DXP604 (Experimental): Part 1A: Single low dose of BGB-DXP604 or placebo; Part 1B: Single high dose of BGB-DXP604 or placebo
  Interventions: Drug: BGB-DXP604; Drug: Placebo
- Part 2 : BGB-DXP604 + BGB-DXP593 (Experimental): Single dose of BGB-DXP593 followed by a single dose of BGB-DXP604 or placebo
  Interventions: Drug: BGB-DXP604; Drug: BGB-DXP593; Drug: Placebo

INTERVENTIONS:
Drug: BGB-DXP604 — Administered as intravenous (IV) infusion over 30 to 60 minutes
Drug: BGB-DXP593 — Administered as intravenous (IV) infusion over 30 to 60 minutes
  Arms: Part 2 : BGB-DXP604 + BGB-DXP593
Drug: Placebo — Placebo to match BGB-DXP593
  Arms: Part 2 : BGB-DXP604 + BGB-DXP593
Drug: Placebo — Placebo to match BGB-DXP604

SUMMARY:
The primary objective of this study is to investigate the safety and tolerability of BGB-DXP604 alone and in combination with BGB-DXP593 in healthy participants

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants are in good general health as determined by the investigator or medically qualified designee, based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
2. Body weight ≥ 50 kg and body mass index (BMI) within the range 18 to 32 kg/m^2 (inclusive)
3. Negative SARS-CoV-2 serology test
4. Negative for COVID-19 based on the nasopharyngeal or oropharyngeal swab with the method of real-time reverse transcription-polymerase chain reaction (rRT-PCR)

Key Exclusion Criteria:

1. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, constituting a risk to the participant when receiving the study drug; or interfering with the interpretation of data
2. Any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that has been resected with no evidence of metastatic disease for 3 years
3. Any history of a severe allergic reaction before enrollment that has a reasonable risk of recurrence during the study
4. Any chronic or clinically significant medical condition that, in the opinion of the investigator, would jeopardize the safety or rights of the participant, including but not limited to type 1 diabetes mellitus, chronic hepatitis; or clinically significant forms of: drug or alcohol abuse, asthma (except for childhood asthma), autoimmune disease, psychiatric disorders, or heart disease
5. Previous receipt of a licensed or investigational biologic agent (such as monoclonal antibodies) within 3 months or 5 half-lives (whichever is longer) before the randomization

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (1):
- Q PHARM, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received normal saline intravenously as placebo at the same volume as BGB-DXP593 or BGB-DXP604
- BGB-DXP604 10 mg/kg: Participants received a single intravenous dose of 10 milligram/kilogram (mg/kg) BGB-DXP604
- BGB-DXP604 30 mg/kg: Participants received a single intravenous dose of 30 mg/kg BGB-DXP604
- BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg: Participants received a single intravenous dose of 15mg/kg of BGB-DXP593 followed by a single intravenous dose of 15mg/kg of BGB-DXP604.
Period: Overall Study
Arm/Group | Placebo | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Started | 6 | 7 | 6 | 6
Completed | 6 | 6 | 6 | 5
Not Completed | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Randomized but Not Treated | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set is defined as all the participants who received either study drug.
Groups:
- BGB-DXP604 10 mg/kg: Participants received a single intravenous dose of 10 mg/kg BGB-DXP604
- Total: Total of all reporting groups
Arm/Group | Placebo | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (12.79) | 28.8 (15.30) | 31.5 (6.98) | 32.2 (11.82) | 30.0 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5 | 3 | 13
  Male | 5 | 2 | 1 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 6 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 0 | 0 | 2
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 5 | 4 | 6 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs)
Description: A TEAE is defined as an adverse event (AE) that had an onset date or a worsening in severity from baseline on or after the administration of study drug and up to 30 days after the dose of study drug.
  An SAE is any untoward medical occurrence that, at any dose results in death, or is life threatening, or requires hospitalization or prolongation of existing hospitalization, or results in disability/incapacity, or is a congenital anomaly/birth defect, or is considered a significant medical AE by the investigator based on medical judgment.
Time Frame: From the day of study drug administration until 30 days after the dose (approximately day 113 )
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Participants with at least 1 TEAE | 5 | 3 | 5 | 6
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 or Higher | 0 | 0 | 0 | 0
  SAE | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Clinically Meaningful Changes in Vital Signs, 12-Lead ECG Parameters and Laboratory Findings
Time Frame: From the day of study drug administration until 30 days after the dose (approximately day 113)
Population: Safety analysis Set
Measure: Number; unit: participants
Arm/Group | Placebo | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants
  Vital Signs | 0 | 0 | 0 | 0
  Laboratory Parameters | 0 | 0 | 0 | 0
  12-Lead ECG Parameters | 0 | 0 | 0 | 0

3. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of BGB-DXP593
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/End of Study (EOS)
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6
μg/mL | 413.4 (52.47)

4. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of BGB-DXP604
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: Pharmacokinetic (PK) Analysis Set included all the participants who received either study drug and had any measurable concentration of study drug(s).
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
μg/mL | 236.9 (38.20) | 744.4 (165.32) | 376.7 (71.14)

5. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast) of BGB-DXP593
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: PK Analysis Set
Measure: Median (Full Range); unit: day*μg/mL
Arm/Group | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6
day*μg/mL | 7282.4 [6329 to 8863]

6. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast) of BGB-DXP604
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: PK Analysis Set
Measure: Median (Full Range); unit: day*μg/mL
Arm/Group | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
day*μg/mL | 5332.3 [4712 to 6456] | 15999.4 [13309 to 22670] | 8850.6 [7227 to 10970]

7. Secondary Outcome: Area Under the Concentration Time Curve From Zero to Infinite Time With Extrapolation of the Terminal Phase(AUCinf) of BGB-DXP593
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: PK Analysis Set
Measure: Median (Full Range); unit: day*μg/mL
Arm/Group | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6
day*μg/mL | 7445.4 [6466 to 9169]

8. Secondary Outcome: Area Under the Concentration Time Curve From Zero to Infinite Time With Extrapolation of the Terminal Phase (AUCinf) of BGB-DXP604
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: PK Analysis Set
Measure: Median (Full Range); unit: day*μg/mL
Arm/Group | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
day*μg/mL | 5801.2 [4984 to 6979] | 17284.1 [14410 to 25171] | 9756.2 [8369 to 12882]

9. Secondary Outcome: Area Under the Concentration Time Curve From Day 1 to Day 29 (AUC0-29) of BGB-DXP593
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22, and 29
Population: PK Analysis Set
Measure: Median (Full Range); unit: day*μg/mL
Arm/Group | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6
day*μg/mL | 4638.0 [3964 to 5227]

10. Secondary Outcome: Area Under the Concentration Time Curve From Day 1 to Day 29 (AUC0-29) of BGB-DXP604
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22, and 29
Population: PK Analysis Set
Measure: Median (Full Range); unit: day*μg/mL
Arm/Group | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
day*μg/mL | 2838.6 [2417 to 3533] | 8282.9 [6811 to 11562] | 4692.8 [4058 to 5754]

11. Secondary Outcome: Time to Achieve Maximum Observed Concentration (Tmax) of BGB-DXP593
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: PK Analysis Set
Measure: Median (Full Range); unit: hours
Arm/Group | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6
hours | 2.93 [2.8 to 8.7]

12. Secondary Outcome: Time to Achieve Maximum Observed Serum Concentration (Tmax) of BGB-DXP604
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: PK Analysis Set
Measure: Median (Full Range); unit: hours
Arm/Group | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
hours | 1.183 [0.97 to 1.25] | 1.167 [1.167 to 6.97] | 1.275 [1.02 to 25.07]

13. Secondary Outcome: Half-life Time (t1/2) of BGB-DXP593
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: PK Analysis Set
Measure: Median (Full Range); unit: day
Arm/Group | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6
day | 20.96 [19.2 to 22.9]

14. Secondary Outcome: Half-life Time (t1/2) of BGB-DXP604
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: PK Analysis Set
Measure: Median (Full Range); unit: day
Arm/Group | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
day | 31.46 [27.3 to 35.6] | 30.56 [27.6 to 33.9] | 32.03 [29.1 to 41.8]

15. Secondary Outcome: Clearance (CL) of BGB-DXP593
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: PK Analysis Set
Measure: Median (Full Range); unit: Liters/day
Arm/Group | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6
Liters/day | 0.15 [0.1 to 0.2]

16. Secondary Outcome: Clearance (CL) of BGB-DXP604
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: PK Analysis Set
Measure: Median (Full Range); unit: Liters/day
Arm/Group | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
Liters/day | 0.11 [0.10 to 0.13] | 0.11 [0.1 to 0.2] | 0.11 [0.1 to 0.2]

17. Secondary Outcome: Volume of Distribution (Vz) of BGB-DXP593
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: PK analysis Set
Measure: Median (Full Range); unit: Liters
Arm/Group | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6
Liters | 4.59 [4.1 to 5.9]

18. Secondary Outcome: Volume of Distribution (Vz) of BGB-DXP604
Time Frame: Day 1 Pre-dose, end of infusion, 6 hours post dose, Days 2,3,4,5,8,15,22,29,43,57,71,85 and 113/EOS
Population: PK Analysis Set
Measure: Median (Full Range); unit: Liters
Arm/Group | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
Liters | 5.00 [4.9 to 5.7] | 4.78 [3.8 to 7.7] | 5.55 [4.6 to 7.0]

19. Secondary Outcome: Clinical Immunogenicity: Number of Participants With Anti-drug Antibodies to BGB-DXP604 and BGB-DXP593
Time Frame: Pre-dose and Days 15,29,57,85 and 113/EOS visit
Population: Anti-drug antibody (ADA) Analysis Set includes all participants who received either study drug and for whom both baseline ADA and ≥ 1 postbaseline ADA results are available
Measure: Number; unit: Percentage of participants
Arm/Group | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
Percentage of participants
  Treatment Induced | 0 | 0 | 0
  Treatment Emergent | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the day of study drug administration until 30 days after the dose (approximately Day 113)
Description: Safety Analysis Set. A TEAE is defined as an AE that had an onset date or a worsening in severity from baseline on or after the administration of study drug and up to 30 days after the dose of study drug.
Arm/Group | Placebo | BGB-DXP604 10 mg/kg | BGB-DXP604 30 mg/kg | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 3/6 | 5/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | BGB-DXP604 10 mg/kg (N=6) | BGB-DXP604 30 mg/kg (N=6) | BGB-DXP593 15 mg/kg + BGB-DXP604 15 mg/kg (N=6)
Headache (Nervous system disorders) | 2 | 2 | 1 | 3
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 0
Catheter site swelling (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT04669262/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT04669262/SAP_001.pdf